CLINICAL TRIAL: NCT02840890
Title: Osteopathy and Prevention of Gastrointestinal Side Effects of the Adjuvant Treatment FEC in Women Treated in Day Hospital for Breast Cancer
Brief Title: Osteopathy and Prevention of Gastrointestinal Side Effects in Women Treated for Breast Cancer
Acronym: PREDIGOSTEO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PREDIGOSTEO
Record Dates: First submitted 2016-04-22; First posted 2016-07-21 (Estimated); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- experimental (Experimental): Patients will have a visceral osteopathic technique perform with continuous pressure on the middle ribs in order to reduce the mechanical stress of the anatomical elements related to liver
  Interventions: Procedure: osteopathic technique
- Placebo (Placebo Comparator): patients will have a relaxing osteopathic technique. A non therapeutic abdominal technique
  Interventions: Procedure: Placebo

INTERVENTIONS:
Procedure: osteopathic technique — Osteopathe will perform continuous pressure on the middle ribs in order to reduce the mechanical stress of the anatomical elements related to liver
  Arms: experimental
Procedure: Placebo — patients will have a relaxing osteopathic technique. A non therapeutic abdominal technique
  Arms: Placebo

SUMMARY:
Adjuvant chemotherapy with the protocol 3 cure of 5-FU + Epirubicine + Cyclophosphamide (FEC100) and 3 cure of Taxotere is a standard treatment in the management of patients with breast cancer and in adjuvant situation.

The efficacy of 3 FEC100 and 3 Taxotere protocol in adjuvant situation for women treated for breast cancer is associated with several invalidating side effects for the quality of life of patients. 92% of women treated will present gastrointestinal toxicities of any grade. 11% will present nausea and vomiting of grade 3-4. Current treatments to prevent these gastrointestinal toxicities include Emend from Day 1 to Day 3 in association with setrons at Day 1 and corticosteroids from Day 1 to Day 3. Despite the marked improvement in gastrointestinal toxicities with preventive treatments, 83% of patients would use alternatives medicine: homeopathy, herbal medicine, acupuncture, hypnotherapy and / or osteopathy.

Osteopathy is a method of care and unconventional therapeutic approach. In France, the professional title of osteopath is recognized. It aims to prevent and treat functional disorders, especially those related to adverse effects of treatment. In oncology, this discipline may have additional support for the patient by limiting the mechanical and physical constraints of sensitive areas to the toxicity of the treatment. In the case of gastrointestinal toxicities of myofascial and musculoskeletal techniques are used in abdominal areas to relieve symptoms. The investigators hypothesis is that osteopathy could have an interest in the management of gastrointestinal toxicities related to chemotherapy in women with breast cancer and in adjuvant treatment situation.

ELIGIBILITY:
Inclusion Criteria:

* Wife
* Age over 18 years
* Operated for a breast cancer stage 1 to 3, in complete resection
* Plan to receive chemotherapy based on FEC100 3 - 3 TAXOTERE
* Nurse Consultation prior to chemotherapy
* planned antiemetic treatment which should include EMEND 125, 80, 80 at J1, J2, J3, ZOPHREN 8 mg IV 1 bulb at J1, Solumedrol 80 mg IV on day 1, Primperan 10 mg 3 tablets a day, from day 1 to day 3, XANAX 0,25 mg 1 tablet morning 1tablet evening from D1 to D3.
* Distance home CGFL 0 to 50 km, 50 to 100 km, 100 to 200 kms.
* Having considered the information note
* written, dated and signed Informed consent

Exclusion Criteria:

* Man
* Metastatic breast cancer
* Breast cancer surgery with incomplete excision
* Digestive disorders known or known digestive disease
* Inability to receive one of the basic elements antibiotic treatment
* Refusal to participate to the trial
* Persons deprived of liberty or under guardianship
* Pregnant woman or likely to be
* Failure to submit to medical testing for geographical reasons (distance home - CGFL more than 200 km), social or psychic
* non-affiliation to a social security scheme or to the State Medical Aid (AME) or the universal medical coverage (CMU)

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2015-11-05 (Actual); Primary Completion 2015-11-05 (Actual); Study Completion 2018-04-20 (Actual)

PRIMARY OUTCOMES:
episode of nausea and / or vomiting | 3 cycles of chemotherapy (each cycle is 21 days for a total of 63 days)

SECONDARY OUTCOMES:
episode of constipation | 3 cycles of chemotherapy (each cycle is 21 days for a total of 63 days)
Quality of life questionnaire(QLQ-C30) | 63 days

CONTACTS AND LOCATIONS:
Overall Officials: Aurélie LAGRANGE, MD, Principal Investigator — Centre Georges François Leclerc
Locations (1):
- CGFL, Dijon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lagrange A, Decoux D, Briot N, Hennequin A, Coudert B, Desmoulins I, Bertaut A. Visceral osteopathic manipulative treatment reduces patient reported digestive toxicities induced by adjuvant chemotherapy in breast cancer: A randomized controlled clinical study. Eur J Obstet Gynecol Reprod Biol. 2019 Oct;241:49-55. doi: 10.1016/j.ejogrb.2019.08.003. Epub 2019 Aug 12. PMID 31430616